CLINICAL TRIAL: NCT05328713
Title: Immune Correlates of Cardiac Structure and Function
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00109701; 1R56HL152803-01 (NIH)
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2022-10

CONDITIONS: Perinatal HIV Infection; Cardiac Fibrosis; Cardiac Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — blood collected for storage for future proteomic profiling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective group with perinatally acquired HIV infection from Duke University Health System clinics
  Interventions: Diagnostic Test: Cardiac MRI
- Control retrospective group: A retrospective age- and sex-matched HIV-uninfected comparator group from Duke University Health System (DUHS) electronic health record (EHR) and imaging database systems

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — This study will use Cardiac MRI to identify subclinical cardiac dysfunction.
  Groups: Prospective group with perinatally acquired HIV infection from Duke University Health System clinics

SUMMARY:
The purpose of this study is to determine the occurrence of scarring of the heart (cardiac fibrosis) and inflammation in those with perinatally acquired Human Immunodeficiency Virus (HIV) infection compared to people not infected with HIV. The information learned from this research may help the investigator to better understand the link between cardiac fibrosis and cardiac dysfunction and inflammation in those with perinatally acquired HIV infection compared to the uninfected.

Participants will have a blood sample, complete a patient questionnaire, and have a Magnetic resonance imaging (MRI) and ultrasound of the heart.

Researchers will review the medical record and past medical history, for information about your heart function and overall health. Research samples and data from this study will be stored indefinitely and used for other research.

There are risks to participate in this study and those risks include side effects from the contrast agent used for the MRI scan, (such as headache and injection site pain), and risks from blood sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 20-45 years of age
2. Willingness and ability to provide signed and dated written informed consent, prior to any study-related procedures
3. Diagnosed with HIV <10 years of age or physician confirmation of perinatal HIV infection
4. On antiretroviral treatment (ART) for at least the last greater than or equal to 6 months
5. Willingness to undergo Cardiovascular magnetic resonance imaging (CMR)
6. Willingness to undergo echocardiogram (ECHO) (may be included if ECHO has been done at Duke in the previous 24 months).
7. Willingness to have research blood draw

Exclusion Criteria:

1. Contraindication to CMR (metal fragments in eyes or face, implanted electronic devices such as pacemakers, defibrillators, cochlear implants, or nerve stimulators, aneurysm clips)
2. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
3. History of anaphylactic reaction to gadolinium contrast
4. Inability to complete an MRI scan in the past due to anxiety
5. Recent acute medical illness resulting in recent hospitalization (in past 90 days)
6. History of: Coronary artery disease (CAD), Myocardial infarction (MI), moderate-severe valvular disease, congenital heart disease, heart failure, non-ischemic CM, Atrial fibrillation/flutter, implantable cardioverter defibrillator (ICD)/pacemaker, myocarditis prior
7. Current Symptoms of Shortness of breath, severe chest pain, palpations, difficulty breathing on exertion, swelling of legs
8. Known to be pregnant or current breastfeeding
9. Known to be on hemodialysis
10. Inability to breath hold for 5-10 seconds
11. Known to have an ejection fraction <45% in the past 24 months
12. Active cancer or cancer chemotherapy or radiation treatment in the prior year.
13. Comorbid inflammatory disease, specifically treated for rheumatoid arthritis (RA) or lupus (SLE)
14. Chronic use of steroids or anti-inflammatory therapy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Recruitment will be from Adult or Pediatric Infectious Disease (ID) Clinics at DUHS and other clinic sites where Duke providers deliver care for HIV.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Myocardial fibrosis by cardiac magnetic resonance (CMR) imaging | Baseline Visit
  Compare myocardial fibrosis for HIV+ and control subjects (unit = percentage)

SECONDARY OUTCOMES:
Cardiac function evaluated using cine cardiac magnetic resonance imaging | Baseline Visit
  Compare Left ventricular ejection fraction (LVEF) for HIV+ and control subjects (unit = percentage) Compare left ventricle (LV) mass for HIV+ and control subjects (unit = grams)
Myocardial edema evaluated using native T2 mapping cardiac magnetic resonance imaging | Baseline Visit
  Compare native T2 mapping values for HIV+ and control subjects (unit = ms)
Diffuse fibrosis evaluated using native T1 mapping cardiac magnetic resonance imaging | Baseline Visit
  Compare native T1 mapping values for HIV+ and control subjects (unit = ms)
Extra-cellular volume (ECV) cardiac magnetic resonance imaging | Baseline Visit
  Compare ECV for HIV+ and control subjects (unit=percentage)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Bloomfield, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams JL, Hung F, Jenista E, Barker P, Chakraborty H, Kim R, McCrary AW, Shah SH, Thielman N, Bloomfield GS. Diffuse myocardial fibrosis is uncommon in people with perinatally acquired human immunodeficiency virus infection. AIDS Res Ther. 2024 Mar 4;21(1):13. doi: 10.1186/s12981-024-00598-4. PMID 38439093